CLINICAL TRIAL: NCT01887691
Title: Sleep Effectiveness and Insulin and Glucose Homeostasis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Melanie Pogach, MD, MMSc, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012P000187
Record Dates: First submitted 2013-06-24; First posted 2013-06-27 (Estimated); Last update posted 2019-12-19 (Actual); Status verified 2018-08

CONDITIONS: Diabetes; Prediabetic; Prediabetes; Glucose Intolerance
Keywords: Diabetes; Prediabetic; Prediabetes; Glucose intolerance; Sleep quality; Continuous glucose monitoring; Diabetes risk; eszopiclone
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; Glucose Intolerance; Sleep Initiation and Maintenance Disorders | interventions — Eszopiclone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- eszopiclone (Experimental): We will evaluate the impact of pharmacologic enhancement of effective sleep with nightly eszopiclone (taken before bedtime for 1 week, home environment) on glycemic profiles (continuous glucose monitoring, 72 hrs) in prediabetics and diabetics compared to pretreatment baseline. The dose of eszopiclone will be the lowest tolerated dose (1-3 mg) via dose escalation and side effect profile assessment.
  Interventions: Drug: eszopiclone

INTERVENTIONS:
Drug: eszopiclone — Eszopiclone at a dose of 1-3 mg (lowest tolerated dose, as determined using a dose escalation schedule and side effect profile)will be taken 30 minutes before bedtime for one week.
  Other Names: Lunesta

SUMMARY:
The purpose of this study is to examine the influence of sleep effectiveness on glucose and insulin metabolism in health and disease (prediabetes and type two diabetes).

We will monitor sleep effectiveness using the sleep spectrogram, obtain serial nocturnal blood glucose and insulin measurements, and assess the impact of pharmacologic enhancement [using eszopiclone (Lunesta), a medication that promotes stable sleep)] on glucose and insulin homeostasis.

We hypothesize that 1: Effective sleep is associated with enhanced insulin sensitivity, relative to ineffective sleep states, and 2: Enhancing sleep effectiveness using eszopiclone (Lunesta) improves 24-hour glucose metabolism in prediabetics and diabetics compared to baseline.

DETAILED DESCRIPTION:
Evidence from experimental studies supports the hypothesis that fragmented or insufficient sleep contributes to impaired glucose and insulin homeostasis. The sleep spectrogram, an EEG-independent measure of sleep effectiveness, maps coupled oscillations of heart rate variability and ECG-derived respiration. In a sample of non-diabetic subjects with and without sleep apnea, we previously explored the association between ECG-spectrogram derived biomarkers and glucose metabolism and found that the marker of effective sleep, High Frequency Coupling (HFC), is associated with reduced diabetes risk (increased Disposition Index). HFC is also enhanced by sedative medications (unpublished data). In this study we will 1.) explore the relationship between sleep effectiveness and insulin sensitivity across the sleep period, by frequently sampling glucose and insulin during nocturnal polysomnography in healthy and prediabetic subjects; and 2.) evaluate the impact of pharmacologic enhancement of effective sleep with nightly eszopiclone (1 week, home environment) on glycemic profiles (continuous glucose monitoring, 72 hrs) in prediabetics and diabetics compared to pretreatment baseline. We expect that desirable glycemic profiles will correlate with the spectrographic marker of effective sleep while undesirable glucose profiles will correlate with the marker of ineffective sleep. Using pharmacologic enhancement of effective sleep, we expect to demonstrate improvement in glycemic profiles in prediabetic and diabetic subjects compared to pre-treatment baseline.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, men and women 18-64 years of age.
* Fluent English speakers.
* Health status as per criteria listed for prediabetes and diabetes (based on 2003 American Diabetes Association criteria and 2009 International Expert Committee Report: Prediabetics will have impaired glucose tolerance with fasting plasma glucose (FPG) 100-125 mg/dL, Hemoglobin A1C 5.7-6.4%, or 2-hour plasma glucose (PG) 140-199 mg/dL after 75-g oral glucose tolerance test (OGTT). Diabetics will have FPG ≥ 126 mg/dL, Hemoglobin A1C ≥ 6.5%, or 2-hour PG ≥ 200 mg/dL on OGTT.

Exclusion Criteria:

* Primary psychiatric disease or conditions which may independently contribute to sleep fragmentation or may hinder the subject's ability to complete the proposed testing:
* Respiratory, liver, or clotting disorders
* History of sleep disordered breathing, Restless legs syndrome or Periodic limb movement disorder or high clinical suspicion of sleep disordered breathing or other sleep disorder (e.g., snoring, excessive daytime sleepiness, frequent napping, excessive motor activity)
* Shift worker or circadian phase disorder
* Abnormal resting ECG, pacemaker, atrial fibrillation or other arrhythmia
* Seizure disorder
* History of depression, bipolar disorder, anxiety disorder, schizophrenia or use of psychiatric medication
* Narcolepsy
* Tobacco or recreational drug use
* Pregnancy or lactation
* Regular use of stimulants or hypnotic medication
* Evidence of sleep apnea (Apnea-Hypopnea Index > 10 on screening sleep study)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2015-08 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
change in continuous glucose profile | comparing 72 hours of baseline and after 1 week of eszopiclone
  continuous glucose monitoring (CGM) results - mean daytime, post prandial and nocturnal glucose between baseline and after 1 week of eszopiclone

SECONDARY OUTCOMES:
change in Sleep effectiveness biomarkers | nightly comparing baseline with post-7 nights of eszopiclone
  M1 results - percentage of high frequency coupling at baseline compared to after 7 nights eszopiclone

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Pogach, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Pogach MS, Punjabi NM, Thomas N, Thomas RJ. Electrocardiogram-based sleep spectrogram measures of sleep stability and glucose disposal in sleep disordered breathing. Sleep. 2012 Jan 1;35(1):139-48. doi: 10.5665/sleep.1604. PMID 22215928